CLINICAL TRIAL: NCT05483218
Title: Evaluation of a Conservative Treatment by Nocturnal Wrist Orthosis in the Non-surgical Management of Carpal Tunnel Syndrome
Brief Title: Evaluation of a Conservative Treatment by Nocturnal Wrist Orthosis in the Non-surgical Management of Carpal Tunnel Syndrome (AMYLYONCARP)
Acronym: ORTHO-2C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO-2C
Record Dates: First submitted 2022-07-05; First posted 2022-08-02 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wrist orthosis (Experimental): group benefiting from an orthosis that supports the wrist by covering the palm of the hand only
  Interventions: Device: Nocturnal wrist orthosis wearing
- wrist-hand-finger orthosis (Experimental): group benefiting from an orthosis that supports the wrist by covering the palm of the hand and the fingers
  Interventions: Device: Nocturnal wrist orthosis wearing

INTERVENTIONS:
Device: Nocturnal wrist orthosis wearing — Nocturnal wearing of one of the 2 wrist orthosis kind

SUMMARY:
This study focuses on the evaluation of 2 nocturnal wrist orthosis prescribed as part of a non-surgical management of carpal tunnel syndrome in order to determine their effectiveness in reducing the symptoms associated with the syndrome and to highlight the superiority or the inferiority of one over the other.

It will also be possible to assess their comfort and compliance as well as the impact of wearing them on neurological and muscular recovery (functional assessment).

DETAILED DESCRIPTION:
After selection of patients suffering from carpal tunnel syndrome during consultation visits, the study will be explained to them, an information sheet and a consent form will be given to them.

A subgroup of patients who have undergone a diagnostic electromyogram at the study center (defined as a functional assessment subgroup) will be randomized independently of the other participants (2 randomization lists will be generated).

The randomization will be done on 2 groups: one benefiting from a wrist orthosis called simple rest, and the other from a wrist-hand-finger orthosis called global rest.

An appointment for making the orthosis will be fixed with the manufacturer within one month of inclusion.

The follow-up will then be done by 2 telephone collection visits at 1 month then at 2 months of the implementation of the device then by a last visit at 3 months consisting in a consultation for the functional assessment subgroup and a phone call for the others.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with unilateral or bilateral, idiopathic or secondary carpal tunnel syndrome, without surgical indication (EMG with myelin sensory signs without axonal involvement)
* signed consent
* Affiliation to social security

Exclusion Criteria:

* Patients with carpal tunnel syndrome with severity criteria
* Patient refusal
* Patient with disorders (psychological, behavioral) that may lead to poor compliance with the study treatment
* Presence of skin lesion in the area of the orthosis
* Current participation in another research protocol involving the human person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Measure and compare the evolution over time of the effectiveness of the 2 nocturnal orthoses | Orthosis implementation, 1 month and 3 months after orthosis implementation
  Score of Boston Carpal Tunnel Syndrome Questionnaire : SEVERITY SCALE OF SYMPTOMS (11 ITEMS): score from 1 to 5 (each item) + FUNCTIONAL EVALUATION SCALE (8 ITEMS): score from 1 to 5 (each item). Higher score means worse outcome.

SECONDARY OUTCOMES:
Evaluate the failure rate of treatment with nocturnal orthosis | 3 months after orthosis implementation
  Need for surgery / infiltration / initiation or increase of anti-inflammatory treatments
Compare the patient's compliance with wearing the 2 types of nocturnal orthosis | 1 month and 3 months after orthosis implementation
  Score of "numerical scale of orthosis wearing duration" : from "never" to "every night". Higher score means better outcome.
Compare the comfort of the 2 types of nocturnal orthosis | 1 month and 3 months after orthosis implementation
  Score of "numerical scale of comfort" : from "1" (very uncomfortable) to "5" (perfectly comfortable). Higher score means better outcome.
Evaluate the impact of the precocity of the conservative treatment on its effectiveness | 1 month and 3 months after orthosis implementation
  Score of Boston Carpal Tunnel Syndrome Questionnaire : SEVERITY SCALE OF SYMPTOMS (11 ITEMS): score from 1 to 5 (each item) + FUNCTIONAL EVALUATION SCALE (8 ITEMS): score from 1 to 5 (each item). Higher score means worse outcome.
Muscle strength recovery | Inclusion and 3 months after orthosis implementation
  For the functional assessment sub-group : measure of muscle strength with a manual dynamometer
Neurological recovery | Inclusion and 3 months after orthosis implementation
  For the functional assessment sub-group : performing of an electromyogram

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Hôpital Neurologique Pierre Wertheimer - Hospices Civils de Lyon, Bron
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Centre Orthopédique Santy, Lyon
  - SELARL de Neurologie Bullukian, Lyon
  - Médipôle Hôpital Mutualiste, Villeurbanne